CLINICAL TRIAL: NCT01884415
Title: Open-label, Phase III, Randomized, Clinical Trial to Evaluate the Efficacy of Two Different Hepatitis B Virus (HBV) Vaccination Schemes in Patients With Hepatic Cirrhosis Candidates to Liver Transplantation
Brief Title: Phase III, Study to Evaluate the Efficacy of Two Different HBV Vaccination Schemes in Patients With Hepatic Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEPATOTRAS
Record Dates: First submitted 2013-06-18; First posted 2013-06-24 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Hepatitis B; Cirrhosis; Awaiting Organ Transplant
MeSH Terms: conditions — Hepatitis B; Fibrosis | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Second HBV vaccination cycle (Experimental): Second cycle of HBV vaccination (0, 1 and 2 months)will be administered. Three intramuscular doses of 40 µg.
  Interventions: Biological: HBV vaccine
- Single dose of HBV vaccine (Active Comparator): Single dose (40µg) of HBV vaccine will be administered at 6 months after 1 cycle of HBV vaccination
  Interventions: Biological: HBV vaccine

INTERVENTIONS:
Biological: HBV vaccine — Patients receive a second cycle of vaccination
  Other Names: HBVAXPRO 40µg HBV vaccine
  Arms: Second HBV vaccination cycle
Biological: HBV vaccine — Patients receive vaccination according to the guidelines.
  Other Names: HBVAXPRO 40µg HBV vaccine
  Arms: Single dose of HBV vaccine

SUMMARY:
The objective of this clinical trial is to compare the response rate obtained with two different vaccination schemes against HBV in cirrhotic patients. These patients must be candidates for liver transplantation, who have failed seroconversion (anti-HBs < 10 IU/ml) after three intramuscular doses of 40 µg.

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhotic patients, potential candidates for liver transplantation, with indication to HBV vaccination (HBsAg negative and anti-HBs negative).
2. Patients under treatment with HBVAXPRO® who do not show a response after the first cycle of vaccination of three intramuscular doses of 40 µg at 0, 1 and 2 months.
3. Patients over 18 years old.
4. Negative pregnancy test.
5. Patients who have given their consent to participate in the study.

Exclusion Criteria:

1. Absolute contraindication to HBV vaccine.
2. Medical history of allergy to any component of the vaccine.
3. Chronic renal failure on hemodialysis.
4. Presence of antibodies against Human Immunodeficiency Virus.
5. Patients with seroconversion (anti-HBs > 10 IU /ml) after the first three doses of vaccine.
6. Lack of consent to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2012-09-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Post-vaccination serological response | At 35 ± 5 days after administration
  To compare the response rate obtained with two different vaccination schemes against HBV in cirrhotic patients potential candidates for liver transplantation, who have failed seroconversion (anti-HBs < 10 IU/ml) after three intramuscular doses of 40 µg at 0, 1 and 2 months.

SECONDARY OUTCOMES:
Association of serological response to HBV vaccination to etiology and severity of cirrhosis | After 6 months
  Etiology and severity of cirrhosis
Association of serological response to HBV vaccination to diabetes presence | After 6 months
  Diabetes
Association of serological response to HBV vaccination to body mass index | At baseline
  Body mass index
Association of serological response to HBV vaccination to anti-Hepatitis B core antigen positive presence | At baseline
  Presence of anti-Hepatitis B core antigen positive
Association of serological response to HBV vaccination to obesity | After 6 months
  Obesity

CONTACTS AND LOCATIONS:
Overall Officials: Juan Manual Pascasio Acevedo, MD, PhD, Study Director — Virgen del Rocío Hospital
Locations (1):
- Virgen del Rocío Hospital, Seville, Spain

REFERENCES:
- [Derived] Giraldez-Gallego A, Rodriguez-Seguel EDP, Valencia-Martin R, Morillo-Garcia A, Salamanca-Rivera C, Ruiz-Perez R, Cuaresma-Duque M, Rosso-Fernandez C, Ferrer-Rios MT, Sousa-Martin JM, Praena-Fernandez JM, Desongles-Corrales T, Rodriguez-Perez A, Camino-Duran F, Gasch-Illescas A, Ampuero-Herrojo J, Pascasio-Acevedo JM. Three double-dose reinforced hepatitis B revaccination scheme for patients with cirrhosis unresponsive to the standard regimen: an open-label randomised clinical trial. Gut. 2023 Dec 7;73(1):166-174. doi: 10.1136/gutjnl-2022-328222. PMID 36963815